CLINICAL TRIAL: NCT04524637
Title: The Utility of Thromboelastography for Predicting the Risk of Coagulation-Related Damages Secondary to Traumatic Brain Injury
Brief Title: The Utility of Thromboelastography in Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, MD, PhD, Associate Professor, Chief Physician, Graduate Supervisor, Shanghai 6th People's Hospital
Other Study IDs: 18PJD034
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injury; Coagulation Disorder
Keywords: Thrombelastography; Coagulation Disorder; Traumatic Brain Injury; Coagulation-related damages
MeSH Terms: conditions — Brain Injuries, Traumatic; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are taken from the antecubital vein for thromboelastography analysis within the first 24 h after head trauma for all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic brain injury: Patients who are delivered within 24 hours after head trauma and sustain isolated traumatic brain injury are included in this study.

SUMMARY:
Hemocoagulation disorder is recognized to have crucial effects on hemorrhagic or ischemic diseases. Coagulation-related damages secondary to traumatic brain injury are common and severe secondary insults of head trauma and often leads to a poor prognosis. In this study, we sought to assess if posttraumatic hemocoagulation disorders determined using thromboelastography are associated with coagulation-related damages secondary to traumatic brain injury, and evaluate their influence on outcome among patients with head trauma. Based on above results, prediction models or risk scoring systems will be further developed and validated to predict coagulation-related damages secondary to traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are delivered to hospital within 24 hours after head trauma
* Patients whose abbreviated injury score (AIS) for other body regions is 3 or less are considered to be isolated traumatic brain injury

Exclusion Criteria:

* Patients with existing prior neurological disease
* Patients with known coagulation disorders
* Patients on anticoagulants and medications known to affect coagulation function within 30 days before trauma
* Patients receiving blood components prior to blood draw
* Patients who deteriorate and die before determining whether coagulation- related damage exists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-80 years old) with isolated traumatic brain injury, who are admitted within 24 hours post-injury are included. To avoid interfering factors, patients with existing prior neurological disease or known coagulation disorders, patients on anticoagulants and medications known to affect coagulation function within 30 days before trauma or receiving blood components prior to blood draw, patients who deteriorate and die before determining whether coagulation-related damage exists are excluded. Clinical data are documented, including age, gender, mechanisms of trauma, types of lesions as evidenced by imaging examination and laboratory examination, etc.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale scores | Six months
  Glasgow Outcome Scale 1 = death; Glasgow Outcome Scale 2 = vegetative state; Glasgow Outcome Scale 3 = severe neurological deficit; Glasgow Outcome Scale 4 = mild neurological deficit and Glasgow Outcome Scale 5 = premorbid level of functioning or completely recovery. Unfavorable outcome is defined as a Glasgow Outcome Scale score of ≤ 3, and favorable outcome is defined as a Glasgow Outcome Scale score of > 3.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, M.D., Ph.D., Study Director — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided